CLINICAL TRIAL: NCT06160739
Title: Role of Sirolimus in Treatment of Microcystic , Mixed Lymphatic and Vascular Malformations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Tarek Ahmed Abd Elsalam, Resident-pediatric surgery department-sohag hospital university, Sohag University
Other Study IDs: soh-Med-23-11-16MS
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Microcystic Lymphatic Malformation; Combined Vascular Malformation; Vascular Malformations
MeSH Terms: conditions — Lymphangioma; Vascular Malformations | interventions — Sirolimus; Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: microcystic & mixed lymphatic malformation
  Interventions: Drug: Sirolimus 1Mg Oral Tablet
- group B: vascular malformation
  Interventions: Drug: Sirolimus 1Mg Oral Tablet

INTERVENTIONS:
Drug: Sirolimus 1Mg Oral Tablet — patients with Microcystic , Mixed Lymphatic and Vascular Malformations will be given sirolimus 1 mg oral tab for 3-6 months with follow up of lesion size by clinical exam & ultrasound & MRI to compare lesion size before & after use of the drug with observation of potential side effects & after exclusion of it before use of the drug

SUMMARY:
Lympho-vascular malformations result from errors in embryologic vasculogenesis involving capillaries, veins, arteries, lymphatics, or a combination of these. Infantile haemangiomas & Vascular malformations like : Capillary malformations & Venous malformations : they increase in size and never regress on their own. & They are generally present at birth, they enlarge in response to infection, hormonal changes or trauma . Lymphatic malformations can be classified into macrocystic (cyst diameter >1cm), microcystic (cyst diameter <1 cm), or mixed , in macrocystic lymphatic malformations, surgery and sclerotherapy are effective . Surgery of microcystic lymphatic malformations remains challenging due to their infiltrative nature & Sclerotherapy is often impossible. As especially large microcystic and mixed malformations are still a therapeutic challenge, pharmaceutical treatment as sirolimus is used in last years as main line of treatment with great efficacy.

DETAILED DESCRIPTION:
Lympho-vascular malformations result from errors in embryologic vasculogenesis involving capillaries, veins, arteries, lymphatics, or a combination of these. Infantile haemangiomas & Vascular malformations like : Capillary malformations & Venous malformations : they increase in size and never regress on their own. & They are generally present at birth, they enlarge in response to infection, hormonal changes or trauma . Lymphatic malformations can be classified into macrocystic (cyst diameter >1cm), microcystic (cyst diameter <1 cm), or mixed , in macrocystic lymphatic malformations, surgery and sclerotherapy are effective . Surgery of microcystic lymphatic malformations remains challenging due to their infiltrative nature & Sclerotherapy is often impossible. As especially large microcystic and mixed malformations are still a therapeutic challenge, pharmaceutical treatment as sirolimus is used in last years as main line of treatment with great efficacy. Sirolimus is a natural macrolide isolated from a bacteria strain of the Streptomyces genus & Streptomyces hygroscopicus . It was initially used as an antibiotic and antifungal agent, subsequent studies have revealed impressive cytostatic, antiproliferative, and immunosuppressive properties . Sirolimus not only prevents the growth of abnormal lymphatics but also induces the partial regression of lesions, without apparent effects on normal lymphatics .

ELIGIBILITY:
Inclusion Criteria:

* from age 6 months to 12 years , not before 6 months to complete their vaccination program & maturation of hepatic enzymes .
* Patients diagnosed with microcystic & mixed Lymphatic malformations .
* After failure of other lines of treatment as regard propranolol , steroid for infantile haemangiomas & Vascular malformations and lymphovascular malformations .
* After failure of surgical excision & injection of bleomycin of Lympho-vascular malformations

Exclusion Criteria:

* Macrocystic Lymphatic malformations & high flow vascular malformations like arterio-venous malformations .
* An active infection that requires systemic treatment during the attack .
* Side effects of the drug as ( history of an allergic reaction to sirolimus or patients who develop severe allergic reaction to drug during treatment , hyperlipidemia , leucopenia , etc… )
* Chronic liver or kidney disease or on chronic drug treatment as (steroids, interferon or chemotherapeutic agents) .
* An immunodeficiency condition such as a human immunodeficiency viral infection or primary immunodeficiency disease.
* Patients who received drug less than 6 months duration .

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * from age 6 months to 12 years , not before 6 months to complete their vaccination program & maturation of hepatic enzymes .
  * Patients diagnosed with microcystic & mixed Lymphatic malformations .
  * After failure of other lines of treatment as regard propranolol , steroid for infantile haemangiomas & Vascular malformations and lymphovascular malformations .
  * After failure of surgical excision & injection of bleomycin of Lympho-vascular malformations
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
changes in size of the lesion | 1 year
  efficacy of sirolimus in decreasing size of the lesion over time , by clinical exam of size lesion & measurement of size of leesion by ultrasound & MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sadick M, Muller-Wille R, Wildgruber M, Wohlgemuth WA. Vascular Anomalies (Part I): Classification and Diagnostics of Vascular Anomalies. Rofo. 2018 Sep;190(9):825-835. doi: 10.1055/a-0620-8925. Epub 2018 Jun 6. PMID 29874693
- [Background] Vlahovic AM, Vlahovic NS, Haxhija EQ. Sirolimus for the Treatment of a Massive Capillary-Lymphatico-Venous Malformation: A Case Report. Pediatrics. 2015 Aug;136(2):e513-6. doi: 10.1542/peds.2014-3469. Epub 2015 Jul 6. PMID 26148957
- [Background] Muller-Wille R, Wildgruber M, Sadick M, Wohlgemuth WA. Vascular Anomalies (Part II): Interventional Therapy of Peripheral Vascular Malformations. Rofo. 2018 Feb 7. doi: 10.1055/s-0044-101266. Online ahead of print. PMID 29415296
- [Background] Adams DM, Wentzel MS. The role of the hematologist/oncologist in the care of patients with vascular anomalies. Pediatr Clin North Am. 2008 Apr;55(2):339-55, viii. doi: 10.1016/j.pcl.2008.01.007. PMID 18381090